CLINICAL TRIAL: NCT06323174
Title: Efficacy and Safety of Co-administered Cagrilintide and Semaglutide (CagriSema) s.c. in Doses 2.4 mg/2.4 mg and 1.0 mg/1.0 mg Once Weekly Versus Placebo in Participants With Type 2 Diabetes Inadequately Controlled on Diet and Exercise
Brief Title: A Research Study to See How Much CagriSema Lowers Blood Sugar and Body Weight Compared to Placebo in People With Type 2 Diabetes Treated With Diet and Exercise
Acronym: REIMAGINE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-4895; 2022-502677-42 (Other: European Medical Agency (EMA)); U1111-1283-0404 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CagriSema Dose 2 (Active Comparator): Participants will receive once-weekly subcutaneous (s.c) injections of CagriSema (cagrilintide and semaglutide) at escalating doses every week in 16-week dose escalation period until target dose (dose 2) of CagriSema (cagrilintide and semaglutide) is achieved and maintained up to 24 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo Dose 2 (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to Cagrisema (cagrilintide and semaglutide) dose 2 for 40 weeks.
  Interventions: Drug: Placebo
- Cagrisema Dose 1 (Active Comparator): Participants will receive once-weekly subcutaneous (s.c) injections of CagriSema (cagrilintide and semaglutide) at escalating doses every week in 8-week dose escalation period until target dose (dose 1) of CagriSema (cagrilintide and semaglutide) is achieved and maintained up to 32 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo Dose 1 (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to Cagrisema (cagrilintide and semaglutide) dose 1 for 40 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive once-weekly cagrilintide subcutaneously.
  Arms: CagriSema Dose 2; Cagrisema Dose 1
Drug: Semaglutide — Participants will receive once-weekly semaglutide subcutaneously.
  Arms: CagriSema Dose 2; Cagrisema Dose 1
Drug: Placebo — Participants will receive placebo matched to cagrilintide and semaglutide subcutaneously.
  Arms: Placebo Dose 1; Placebo Dose 2

SUMMARY:
This study will look at how much CagriSema helps participants with type 2 diabetes lower their blood sugar and body weight. CagriSema is a new investigational medicine. Doctors may not yet prescribe CagriSema. CagriSema will be compared to a "dummy" medicine (also called "placebo") that has no effect on the body. Participants will get either CagriSema or "dummy" medicine. Which treatment participants get is decided by chance. For each participant, the study will last for about one year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 years or above at the time of signing the informed consent
* Diagnosed with type 2 diabetes >=30 days before screening
* HbA1c 7.0-9.5 percent (53-80 millimoles per mole [mmol/mol]) (both inclusive) as determined by central laboratory at screening
* Body mass index (BMI) >=23 kilograms per square meter (kg/m^2) at screening. BMI will be calculated in the electronic case report form (eCRF) based on height and body weight at screening

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method
* Renal impairment with estimated Glomerular Filtration Rate less than 30 milliliter per minute per 1.73 square meter (ml/min/1.73 m^2) as determined by central laboratory at screening
* Treatment with any medication for the indication of diabetes or obesity within 90 days before screening. However, short term insulin treatment for a maximum of 14 consecutive days and prior insulin treatment for gestational diabetes are allowed
* History of use of any injectable therapy for diabetes or obesity. However, short term insulin treatment for a maximum of 14 consecutive days and prior insulin treatment for gestational diabetes are allowed
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 40)
  Measured as percentage (%)-points.

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 40)
  Measured in %.
Number of participants who achieve greater than or equal to (>=) 10% body weight reduction | From baseline (week 0) to end of treatment (week 40)
  Measured as count of participants.
Number of participants who achieve >=15% body weight reduction | From baseline (week 0) to end of treatment (week 40)
  Measured as count of participants.
Number of participants who achieve HbA1c target values of less than (<) 7.0% (<53 millimoles per mole [mmol/mol]) | At end of treatment (week 40)
  Measured as count of participants.
Number of participants who achieve HbA1c target values of less than or equal to (<=) 6.5% (<= 48 mmol/mol) | At end of treatment (week 40)
  Measured as count of participants.
Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of treatment (week 40)
  Measured in millimoles per liter (mmol/L).
Number of participants who achieve >=5% body weight reduction | From baseline (week 0) to end of treatment (week 40)
  Measured as count of participants.
Number of participants who achieve >=20% body weight reduction | From baseline (week 0) to end of treatment (week 40)
  Measured as count of participants.
Change in waist circumference | From baseline (week 0) to end of treatment (week 40)
  Measured in centimeters (cm).
Change in systolic blood pressure (SBP) | From baseline (week 0) to end of treatment (week 40)
  Measured in millimeters of mercury (mmHg).
Change in diastolic blood pressure (DBP) | From baseline (week 0) to end of treatment (week 40)
  Measured in mmHg.
Ratio to baseline in high sensitivity C-reactive protein (hsCRP) | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Ratio to baseline in lipids: Total cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Ratio to baseline in lipids: High-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Ratio to baseline in lipids: Low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Ratio to baseline in lipids: Very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Ratio to baseline in lipids: Triglycerides | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Ratio to baseline in lipids: Free fatty acids | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Ratio to baseline in lipids: Non-HDL cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Number of participants who achieve type 2 diabetes (T2D) remission (HbA1c <6.5% and no antidiabetic medication) | At end of study (week 52)
  Measured as count of participants.
Ratio to baseline in oral glucose tolerance test (OGTT) based oral glucose disposition index (DIo) | From baseline (week 0) to end of treatment (week 40)
  Measured as ratio.
Change in experienced level of energy as measured by the SF-36v2 Health Survey Acute (SF-36v2) Vitality score | From baseline (week 0) to end of treatment (week 40)
  Measured as score points. SF-36v2 Acute measures Health-Related Quality of Life (HRQoL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10.
  Higher scores indicate better functional health and well-being. The vitality score range is from 25.6 to 69.1.
Change in SF-36v2 score: Physical Component Summary score | From baseline (week 0) to end of treatment (week 40)
  Measured as score points. SF-36v2 Acute measures HRQoL. The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The score range for physical component summary is 6.1 to 79.7.
Change in SF-36v2 score: Mental Component Summary score | From baseline (week 0) to end of treatment (week 40)
  Measured as score points. SF-36v2 Acute measures HRQoL. The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The score range for mental component summary score is -3.8 to 78.7.
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) score | From baseline (week 0) to end of treatment (week 40)
  Measured as score points. DTSQs measures treatment satisfaction and diabetes-specific quality of life. The measure consists of 8 items yielding 1 global score and 2 single item scores. Higher scores on the global score indicate greater satisfaction with treatment. Lower scores on the single-item scores indicate BG levels closer to the ideal, while higher scores indicate problems. Single-item scores (score range): Perceived frequency of hyperglycaemia (0-6), Perceived frequency of hypoglycaemia (0-6). Global score (score range): Total Treatment Satisfaction (0-36).
Change in leptin | From baseline (week 0) to end of treatment (week 40)
  Measured in nanograms per milliliter (ng/mL).
Change in soluble leptin receptor | From baseline (week 0) to end of treatment (week 40)
  Measured in ng/mL.
Number of Treatment Emergent Adverse Events (TEAEs) | From baseline (week 0) to end of treatment +7 weeks (week 47)
  Measured as count of events.
Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol (54 milligrams per deciliter [mg/dL]), confirmed by blood glucose (BG) meter | From baseline (week 0) to end of treatment +7 weeks (week 47)
  Measured as count of episodes.
Number of severe hypoglycaemic episodes (level 3): hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold | From baseline (week 0) to end of treatment + 7 weeks (week 47)
  Measured as count of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (50):
- United States (21):
  - Nat Res Inst Huntington Park, Huntington Park, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Southern California Dermatology, Santa Ana, California
  - Encore Medical Research LLC, Hollywood, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Encore Medical Research of Weston, Weston, Florida
  - Alliance for Multispec Res, Newton, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Arcturus HC PLC Troy Med Res, Troy, Michigan
  - Southgate Medical Group, LLP, West Seneca, New York
  - Summit Research Network Oregon Inc., Portland, Oregon
  - Holston Medical Group, Kingsport, Tennessee
  - Amarillo Medical Specialists, Amarillo, Texas
  - Elligo Clin Res Centre, Austin, Texas
  - Headlands Research Brownsville, Brownsville, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Northeast Clinical Research of San Antonio, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Sugar Lakes Family Practice PA, Sugar Land, Texas
  - Valley Diab. & Endo Comp Ctr, Weslaco, Texas
  - TPMG Clinical Research, Newport News, Virginia
- China (5):
  - Chinese People's Liberation Army General Hospital-Endocrinology, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Nanjing Medical University-Endocrinology, Nanjing, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Ji'Nan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
- Hungary (4):
  - Belinus Bt., Debrecen, Hajdú-Bihar
  - Borbánya Praxis E.Ü. Kft., Nyíregyháza, Szabolcs-Szatmar Varmegye
  - Szent Margit Rendelőintézet Nonprofit Kft., Budapest
  - PVN Kutato Kft., Budapest
- Italy (4):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Policlinico Mater Domini Università di Catanzaro, Catanzaro
  - IRCCS Ospedale San Raffaele Milano, Milan
  - Azienda Ospealiero Universitaria Policlinico Umberto I, Roma
- Poland (7):
  - Centrum Medyczne Medyk Sp. z o.o., Rzeszów, Podkarpackie Voivodeship
  - Osteo-Medic s.c. A. Racewicz, J. Supronik, Bialystok
  - Renew Clinic Sp. z o.o., Bialystok
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - NBR Polska Tomasz Klodawski, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
  - Velocity Nova Sp. z o.o., Zamość
- Saudi Arabia (5):
  - King Abdulaziz Hospital-Al Ahsa-National Guard, Al Ahsa
  - National Guard Hospital - Jeddah, Jeddah
  - King Fahad Medical City, Riyadh
  - King Khaled University Hospital,King Saud Univ. Med. City, Riyadh
  - King Salman Bin Abdulaziz Hospital, Riyadh
- Serbia (4):
  - CHC Zvezdara, Clinical department for endocrinology, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Policlinic for diabetes, Zaječar

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com